CLINICAL TRIAL: NCT02191592
Title: Identification of Unique Tinnitus Subgroups Using Ecological Momentary Assessment (EMA).
Brief Title: EMA-Defined Tinnitus Subgroups
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine
Other Study IDs: 201407024
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Tinnitus
Keywords: Tinnitus; EMA; Bothersome
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to test a new way of measuring the severity of tinnitus using a tool called Ecological Momentary Assessment (EMA) of Tinnitus. We will compare the relationship with this tool with another widely used questionnaire. Previous studies we have done suggest there are different patterns of tinnitus bother; we plan to explore how often these patterns occur, and how many patterns of tinnitus bother there are. And lastly we want to test how reliable this type of testing is for measuring the amount of bother people experience from their tinnitus.

Hypothesis 1: We will be able to identify 6 or more distinctive patterns of tinnitus.

Hypothesis 2: EMA will provide a reliable method for more accurately capturing the amount of bother individuals have from tinnitus.

DETAILED DESCRIPTION:
You to need to complete this brief survey to determine if you meet the criteria for participation in the study. You are free to skip any questions that you prefer not to answer. We will only use the information you provide in this survey to determine if you qualify for the EMA-Defined Tinnitus Subgroups study.

To be in this study, you will be required to have a smart phone that can receive text messages, is connected to the internet, and will allow you to connect via the internet to a Washington University secure server. It is necessary to connect to the Washington University server in order to complete a short survey four times a day for two separate two-week periods.

The study involves us sending you text messages at 4 random times during the day, between the hours of 8: 00 am - 9: 00 pm. The texts prompt you to click on a link and respond to a short EMA survey regarding what you are doing, what your environment is, and how your tinnitus is at that moment. These text messages will be sent daily for two weeks. Then you will have two weeks off. Finally you will again receive the text messages asking for you to respond to the survey for two more weeks. You will receive a total of 112 text messages over four weeks. In addition we will send you four emails or texts asking you to complete a survey at the following times: before you complete your first set of EMA surveys, at the end of the first set EMA surveys, prior to starting the second set of EMA surveys, and a final time after you have completed the final EMA survey. This study requires no visits to Washington University.

In order to participate you must complete this short prescreening survey to see if you qualify.

ELIGIBILITY:
Inclusion Criteria:

* Age between the ages of 21 and 80.
* Have subjective, unilateral or bilateral, tinnitus of 6 months' duration or longer.
* Must be score of 1, 2, 3, or 4 on Global Bother Score. (Range is 0-4, with 0 being not bothered and 4 being extremely bothered)
* Must have access to a smart phone device compatible with the notification system.
* Must be able to read, write, and understand English.

Exclusion Criteria:

* Tinnitus related to Workman's Compensation Claim or other litigation-related situations.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from Otolaryngology Clinics and from Tinnitus Support Groups
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Ecological Momentary Assessment of Tinnitus | Week 1-2 and Week 4-6
  This is a two week period of capturing real time data regarding a subjects tinnitus bother, environment, and activity at random periods of the day. This is a patient self report measure, but captures data in real time vs. asking them to recall information retrospectively.

SECONDARY OUTCOMES:
Tinnitus Functional Index (TFI) | Pre-Screening, Baseline, Week 2, Week 4, Week 6
  This is a retrospective patient self-report questionnaire. It scores the severity of patient bother experienced from their tinnitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Stone AA, Shiffman S. Capturing momentary, self-report data: a proposal for reporting guidelines. Ann Behav Med. 2002 Summer;24(3):236-43. doi: 10.1207/S15324796ABM2403_09. PMID 12173681
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Freedman MJ, Lester KM, McNamara C, Milby JB, Schumacher JE. Cell phones for ecological momentary assessment with cocaine-addicted homeless patients in treatment. J Subst Abuse Treat. 2006 Mar;30(2):105-11. doi: 10.1016/j.jsat.2005.10.005. PMID 16490673
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Stone AA, Schwartz JE, Broderick JE, Shiffman SS. Variability of momentary pain predicts recall of weekly pain: a consequence of the peak (or salience) memory heuristic. Pers Soc Psychol Bull. 2005 Oct;31(10):1340-6. doi: 10.1177/0146167205275615. PMID 16143666
- [Background] Axelsson A, Ringdahl A. Tinnitus--a study of its prevalence and characteristics. Br J Audiol. 1989 Feb;23(1):53-62. doi: 10.3109/03005368909077819. PMID 2784987
- See also: Clinical Outcomes Research Office Web-site — http://otooutcomes.wustl.edu